CLINICAL TRIAL: NCT03677466
Title: Clinical Trial Appreciating Intramyocardial Haemorrhage in Patients With Primary STEMI and Different Reperfusion Strategies (Pharmaco Invasive Strategy and Primary PCI)
Brief Title: Intramyocardial Haemorrhage in Patients With Primary STEMI
Acronym: HaemInCor
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tomsk National Research Medical Center of the Russian Academy of Sciences (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: HaemInCor
Record Dates: First submitted 2018-09-17; First posted 2018-09-19 (Actual); Last update posted 2019-04-05 (Actual); Status verified 2019-03

CONDITIONS: Myocardial Infarction; STEMI; Myocardial Necrosis; Myocardial Injury
Keywords: Intramyocardial haemorrhage; Myocardial Infarction; ST Elevation Myocardial Infarction; Primary Percutaneous Coronary Intervention; Pharmaco invasive strategy; Fibrinolytic therapy; Global longitudinal strain; Myocardial Necrosis; Coronary Artery Disease
MeSH Terms: conditions — Myocardial Infarction; ST Elevation Myocardial Infarction; Coronary Artery Disease | interventions — Tenecteplase; Tissue Plasminogen Activator; Streptokinase

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pharmaco-invasive strategy (Experimental): Fibrinolytic therapy (Streptokinase, Alteplasa, Tenecteplasa in standard dose) is conducted within 12 h of symptom onset in the pre-hospital setting if primary PCI cannot be performed within 120 min from STEMI diagnosis. Then PCI is performed to all of patients.
  Interventions: Drug: Pharmaco-invasive strategy
- Primary PCI (Active Comparator): Primary percutaneous coronary intervention (PCI) in patients with primary STEMI
  Interventions: Procedure: Primary PCI

INTERVENTIONS:
Drug: Pharmaco-invasive strategy — Patient with primary STEMI will received standard doses of fibrinolytics with following PCI.
  After reperfusion strategies will be conducted cardiovascular magnetic resonance (CMR) imaging with contrast (Gadovist) in regime inversion recovery time, regime T-2 weighted images, T1-weighted images. and Global Longitudinal Strain measured with echocardiography.
  Other Names: Metalyse; Actilyse; Tenecteplase; Alteplase; Streptokinase
  Arms: Pharmaco-invasive strategy
Procedure: Primary PCI — After primary PCI patients will be conducted cardiovascular magnetic resonance (CMR) imaging with contrast (Gadovist) in regime inversion recovery time, regime T-2 weighted images, T1-weighted images and Global Longitudinal Strain measured with echocardiography.
  Arms: Primary PCI

SUMMARY:
The purpose of the study is to assess the frequency and intensity of intramyocardial haemorrhage in patients with primary STEMI and different reperfusion strategies.

DETAILED DESCRIPTION:
The study non-randomized, opened, controlled. In half of patients despite on carried in-time reperfusion therapy intramyocardial haemorrhage determined after a long-term period of severe ischemia. Earlier, definition of intramyocardial haemorrhage was possible only by autopsy. Nowaday, cardiac contrast MRI is the best diagnostic method, which allows to assess the regional and global function of the LV, structural changes in myocardial tissue and also in T2 mode it became assessable to reveal intramyocardial haemorrhage.

Taking into account the results of previous researches, it can be concluded that the intramyocardial haemorrhage was determined in half of patients with primary PCI [1]. An influence of fibrinolytic therapy to the intramyocardial haemorrhage was conducted in small group of patients in one trial, and therefore further data will be actual and useful [2].

It is planned to study 60 patients with primary STEMI using standard therapy. The patients will be divided into 2 groups. Patients of the 1st group will be treated by pharmaco-invasive strategy. The 2nd group will be treated by primary PCI. Patients in all groups after reperfusion strategies will be conducted cardiac contrast MRI for detection intramyocardial haemorrhage within 2 days onset. At day 7 and through 3 months, the clinical condition of the patients will be assessed and cardiac ultrasound will be performed for the evaluation of myocardial contractile function and 2D global longitudinal strain. Also, the incidence rate of secondary endpoints will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years at time of randomization (18 years and older);
* Acute myocardial infarction;
* Reperfusion of the infarct-related coronary artery in terms within 12 h of symptom onset;
* Written the informed consent to participate in research;

Exclusion Criteria:

* Inability to obtain informed consent;
* Patients previously undergone endovascular / surgical revascularization of coronary artery;
* Severe comorbidity;
* History of myocardial infarction;
* History of intracranial haemorrhage;
* Pulmonary edema, cardiogenic shock;
* Creatinine clearance <30 mL/min or dialysis;
* Unable to undergo or contra-indications for MRI;
* Allergy for contrast agent;
* Indication or use of oral anticoagulant therapy;
* Major bleedind;
* Atrio-ventricular block II and III degree;
* Active gastroduodenal ulcer;
* Aortic dissection;
* Acute psychotic disorders

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2018-01-25 (Actual); Primary Completion 2018-10-30 (Actual); Study Completion 2019-03-20 (Actual)

PRIMARY OUTCOMES:
Intramyocardial haemorrhage in primary STEMI measure | 2 days
  Intramyocardial haemorrhage (%) in patients with primary STEMI as assessed by cardiac magnetic resonance imaging 2 days after reperfusion

SECONDARY OUTCOMES:
Left ventricular ejection fraction (LVEF) recovery measure | 3 months (with intermediate measurement at day 7 after reperfusion)
  Left ventricular ejection fraction (LVEF) (%) recovery measured with echocardiography 7 days and 3 months after reperfusion strategies
Global Longitudinal Strain | 3 months (with intermediate measurement at day 7 after reperfusion)
  Global Longitudinal Strain (%) measured with echocardiography 7 days and 3 months after reperfusion strategies
Recurrent myocardial infarction measure | 3 months
  Incidence of recurrent myocardial infarction (%) 3 months after STEMI
Heart failure incidence measure | 3 months
  Incidence of heart failure (%) 3 months after STEMI
Stroke incidence measure | 3 months
  Incidence of stroke (%) 3 months after STEMI
Mortality measure | 3 months
  Mortality rate (%) 3 months after STEMI
Major bleeding incidence measure | 3 months
  Incidence of major bleeding (%) 3 months after STEMI

CONTACTS AND LOCATIONS:
Overall Officials: Evgeny V. Vyshlov, Principal Investigator — Tomsk NRMC
Locations (1):
- Cardiology Research Institute, Tomsk, Russia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Hamirani YS, Wong A, Kramer CM, Salerno M. Effect of microvascular obstruction and intramyocardial hemorrhage by CMR on LV remodeling and outcomes after myocardial infarction: a systematic review and meta-analysis. JACC Cardiovasc Imaging. 2014 Sep;7(9):940-52. doi: 10.1016/j.jcmg.2014.06.012. PMID 25212800
- [Result] Carrick D, Haig C, Ahmed N, McEntegart M, Petrie MC, Eteiba H, Hood S, Watkins S, Lindsay MM, Davie A, Mahrous A, Mordi I, Rauhalammi S, Sattar N, Welsh P, Radjenovic A, Ford I, Oldroyd KG, Berry C. Myocardial Hemorrhage After Acute Reperfused ST-Segment-Elevation Myocardial Infarction: Relation to Microvascular Obstruction and Prognostic Significance. Circ Cardiovasc Imaging. 2016 Jan;9(1):e004148. doi: 10.1161/CIRCIMAGING.115.004148. PMID 26763281